CLINICAL TRIAL: NCT04637230
Title: Prevention of Stroke and Sudden Cardiac Death by Recording of 1-Channel Electrocardiograms
Acronym: PRICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: A-Rhythmik GmbH (Other)
Responsible Party: Sponsor
Organization: Lanserhof (Other)
Other Study IDs: 20-139
Record Dates: First submitted 2020-11-17; First posted 2020-11-19 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Sinus Rhythm; Atrial Fibrillation; Atrial Premature Complexes; Ventricular Premature Complexes; Ventricular Tachycardia, Nonsustained
Keywords: Automated ECG diagnosis
MeSH Terms: conditions — Atrial Fibrillation; Atrial Premature Complexes; Ventricular Premature Complexes; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Sinus Rhythm: Subjects/patients in normal sinus rhythm
  Interventions: Diagnostic Test: Electrocardiogram analysis by Artificial Intelligence
- Atrial Fibrillation: Patients with atrial fibrillation
  Interventions: Diagnostic Test: Electrocardiogram analysis by Artificial Intelligence
- Atrial Premature Complexes: Patients with atrial premature complexes in between sinus beats
  Interventions: Diagnostic Test: Electrocardiogram analysis by Artificial Intelligence
- Ventricular Premature Complexes: Patients with ventricular premature complexes in between sinus beats
  Interventions: Diagnostic Test: Electrocardiogram analysis by Artificial Intelligence
- Ventricular Tachycardia, Nonsustained: Patients with episodes of nonsustained ventricular tachycardia in between sinus beats
  Interventions: Diagnostic Test: Electrocardiogram analysis by Artificial Intelligence

INTERVENTIONS:
Diagnostic Test: Electrocardiogram analysis by Artificial Intelligence — 1-channel electrocardiograms are collected to train an Artificial Intelligence in the automatic diagnosis of regular and irregular heart rhythms

SUMMARY:
Single-channel electrocardiograms (lead I of 12-lead surface ECG; 30 seconds) will be collected from subjects/patients at 11 clinical centers in Germany to train an Artificial Intelligence in the automatic diagnosis of regular and irregular heart rhythms. Heart rhythms of interest are normal sinus rhythm (SR), atrial fibrillation (AF), atrial premature beats (APBs), ventricular premature beats (VPBs), and nonsustained ventricular tachycardia (VT). Per diagnosis, 20,000 ECGs are required, for a total of 100,000 ECGs to be obtained from approximately 10,000 subjects/patients.

DETAILED DESCRIPTION:
In phase 1 of a research project titled 'Prevention of stroke and sudden cardiac death by Recording of 1-Channel Electrocardiograms' (PRICE), a total of 100,000 30-sec single-channel ECGs (lead I of 12-lead surface ECG) will be collected from approximately 10,000 subjects/patients at 11 participating clinical centers in Germany. Relevant baseline clinical patient characteristics will also be recorded. The ECGs, diagnosed by an experienced electrophysiologist (diagnostic gold standard), will be fed into an Artificial Intelligence (AI) for the automatic detection of normal sinus rhythm (SR), atrial fibrillation (AF), atrial premature beats (APBs), ventricular premature beats (VPBs), and nonsustained ventricular tachycardia (VT). It is expected that the overall diagnostic accuracy of the AI against an experienced electrophysiologist will be on the order of 95%.

In PRICE phase 2, ECG diagnosis by the AI will be compared with the diagnosis by 3 general cardiologists of the same ECGs. It is expected that the AI will surpass the general cardiologists in terms of diagnostic accuracy.

The final clinical phase of the PRICE project will comprise a randomized controlled community trial of risk patients to establish the superiority in stroke prevention of AI detection of AF on smart-watch ECGs vs. no AF detection.

ELIGIBILITY:
Inclusion Criteria:

* Heart rhythm of interest present on ECG

Exclusion Criteria:

* Patient incapable of or not willing to sign informed consent form

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from tertiary care centers
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of AI | 1 year
  Overall diagnostic accuracy of the AI in the diagnosis of normal SR, AF, APBs, VPBs, and nonsustained VT (gold standard: diagnosis by experienced electrophysiologist)
ECG R-R interval | Immediate
  30-sec mean and standard deviation of R-R intervals
ECG QRS-complex duration | Immediate
  Measurement of width/duration of QRS complex; distinction between "narrow" (<=110ms) and "wide" (>110ms)
ECG QRS-complex fragmentation | Immediate
  Assessment of presence ("Yes") or absence ("No") of QRS-complex fragmentation
ECG QTc interval | Immediate
  Calculation of heart rate corrected QT interval (QTc) via Bazett formula from measured QT interval
ECG T wave inversion | Immediate
  Assessment of presence ("Yes") or absence ("No") of T wave inversion

SECONDARY OUTCOMES:
ECG P wave | Immediate
  Assessment of presence ("Yes") or absence ("No") of P wave on ECG; measurement of P-wave duration (in ms)
ECG PQ interval | Immediate
  Measurement of PQ interval (onset of P wave to onset of Q wave) on ECG
ECG QT interval | Immediate
  Measurement of QT interval (onset of Q wave to end of T wave) on ECG

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, MD, Principal Investigator — Universitäres Herzzentrum, Lübeck, Germany
Locations (1):
- Universitäres Herzzentrum, Lübeck, Germany, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: No